CLINICAL TRIAL: NCT01700062
Title: Assessment the Effect of Medium-Calorie TPN on Patients With Gastrointestinal Cancer Undergoing Surgery
Brief Title: Medium Calorie Parenteral Nutrition on Patients With Gastrointestinal Cancer Undergoing Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, JUI-FEN CHUANG, Department of pharmacy, leader, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KMUH-IRB-960022
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Neoplasms
Keywords: medium-calorie; standard calorie; parenteral nutrition
MeSH Terms: conditions — Colorectal Neoplasms; Hyperphagia | interventions — Parenteral Nutrition, Total

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medium calorie (Experimental)
  Interventions: Dietary Supplement: Total Parenteral Nutrition (TPN)
- standard calorie (Experimental)
  Interventions: Dietary Supplement: Total Parenteral Nutrition (TPN)

INTERVENTIONS:
Dietary Supplement: Total Parenteral Nutrition (TPN) — Medium calorie ,Nonprotein calories 20 Kcal/Kg/day,Protein 1g/Kg,Fat emulsion 0.5 g/kg/day D1-D6 post OP standard calorie, Nonprotein calories 30 Kcal/Kg/day,Protein 1.5 g/Kg,Fat emulsion 50g/day D1-D6 post OP

SUMMARY:
aimed at investigating the efficacy, safety, and clinical outcome of Medium-Calorie or standard-calorie total parenteral nutrition (TPN) for patients with gastrointestinal cancer undergoing surgery

DETAILED DESCRIPTION:
biochemistry data Various inflammation-related cytokines clinical outcome hospital stay

ELIGIBILITY:
Inclusion Criteria:

* Patients considered for major surgery for colorectal cancer Expected requirement for post operative PN or TPN of at least for 7 days Age >18 Hemodynamically stable Written Informed Consent

Exclusion Criteria:

* Hemodynamic failure of any organ Renal insufficiency Patients with severe liver dysfunction Albumin < 3g/dL DM with poor blood sugar control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
biochemistry data; Various inflammation-related cytokines ; | 7 days

SECONDARY OUTCOMES:
clinical outcome(hospital stay..) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: JF CHUANG, M.S., Principal Investigator — Department of pharmacy, Kaohsiung Medical University Hospital, Kaohsiung, Taiwan; JY WANG, M.D., Study Chair — Departments of Surgery Kaohsiung Medical University Hospital, Kaohsiung, Taiwan; YB HUANG, Ph.D., Study Director — Departments of Pharmacy, Kaohsiung Medical University Hospital, Kaohsiung, Taiwan
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Kaohsiung, Taiwan